CLINICAL TRIAL: NCT02809053
Title: A Randomized, Double-blind, Multi-center, Multi-national Trial to Evaluate the Efficacy, Safety, and Immunogenicity of SAIT101 Versus Rituximab as a First-line Immunotherapy Treatment in Patients With Low Tumor Burden Follicular Lymphoma
Acronym: RAMO-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Archigen Biotech Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGB002
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Lymphoma, Follicular
Keywords: low tumor burden follicular lymphoma (LTBFL)
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAIT101 (Experimental)
  Interventions: Biological: SAIT101
- MabThera® (Active Comparator)
  Interventions: Biological: MabThera®

INTERVENTIONS:
Biological: SAIT101 — Dose of 375mg/m2 body surface area (BSA) i.v. on Days 1, 8, 15, and 22
  Arms: SAIT101
Biological: MabThera® — Dose of 375mg/m2 body surface area (BSA) i.v. on Days 1, 8, 15, and 22
  Other Names: Rituximab
  Arms: MabThera®

SUMMARY:
This is a Randomized, Double-blind, Multi-center, Multi-national Trial to Evaluate the statistical equivalence of efficacy, safety and immunogenicity of SAIT101 Versus Rituximab as a First-line Immunotherapy Treatment in asymptomatic patients with Low Tumor Burden Follicular Lymphoma.

DETAILED DESCRIPTION:
This is a Randomized, Double-blind, Multi-center, Multi-national Trial to Evaluate the statistical equivalence of efficacy, safety and immunogenicity of SAIT101 Versus Rituximab as a First-line Immunotherapy Treatment in asymptomatic patients with Low Tumor Burden Follicular Lymphoma. Patients will be randomized in a 1:1 ratio to receive study drug once a week for 4 weeks, and will then be followed up for up to 52 weeks after the first dose. Randomization will be stratified by inclusion in the PK/PD sub-population and Follicular lymphoma international prognostic index 2 (FLIPI-2) score.

Visits are scheduled at Weeks 1, 2, 3, and 4 (study drug infusion visits), and then at Weeks 5, 12, 20, 28, 36, and 52 (i.e., End of Study [EOS]). Efficacy response assessments will be performed at Weeks 12 and 28, while safety assessments will continue until end of Study (EOS).

The primary objectives is to compare the efficacy of SAIT101 with rituximab licensed in the European Union (hereafter designated MabThera®, brand name in EU) when administered as a first-line immunotherapy in patients with low tumor burden follicular lymphoma (LTBFL) and the secondary objectives is to evaluate SAIT101 versus MabThera® with respect to safety and tolerability, immunogenicity and Pharmacokinetics (PK)/Pharmacodynamics (PD) in a sub-population of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-confirmed Low Tumor Burden Follicular Lymphoma, without B symptoms, Ann Arbor stage II to Non-Hodgkin's Lymphoma (NHL) (CD20+ Follicular Lymphoma of Grades 1, 2, or 3a)
2. Low tumor burden according to The Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria defined as:

   * Normal serum lactate dehydrogenase (LDH)
   * No mass ≥7 cm.
   * Less than 3 nodal sites, each with diameter >3 cm
   * No systemic or B symptoms (fever >38°C for 3 consecutive days; recurrent, drenching night sweats; unintentional weight loss exceeding 10% body weight in the last 6 months.
   * No splenomegaly ≥16 cm by CT scan.
   * No risk of vital organ compression.
   * No pleural or peritoneal serous effusion.
   * No leukemic phase >5,000/µL circulating tumor cells.
   * No cytopenias (defined as platelets <100,000/mm3, hemoglobin <10 g/dL, or absolute neutrophil count <1,500/mm3).
3. Patients not previously treated for their FL, including any previous treatment for FL under clinical trials except localized radiation therapy for previous limited stage disease.

Exclusion Criteria:

1. Previous treatment with any chemotherapy and/or rituximab or other monoclonal antibody.
2. Prior radiotherapy completed <28 days before study enrollment.
3. Anticipated need for concomitant administration of any other experimental drug, or a concomitant chemotherapy, anticancer hormonal therapy, radiotherapy, or immunotherapy during study participation.
4. Concomitant disease which requires continuous therapy with corticosteroids at doses equivalent to prednisolone >20 mg/day.
5. Transformation to high-grade lymphoma secondary to previously untreated low-grade lymphoma.
6. Prior or concomitant malignancies within 5 years prior to screening, with the exceptions of non-melanoma skin cancer, adequately treated carcinoma in situ of the cervix, adequately treated breast cancer in situ, and localized prostate cancer stage T1c, provided that the patient underwent curative treatment and remains relapse free.
7. Patients with a body surface area >3.0 m2.
8. Major surgery (excluding lymph node biopsy) within 28 days prior to randomization.
9. Primary or secondary immunodeficiency (history of, or currently active), including known history of human immunodeficiency virus (HIV) infection or positive test at screening.
10. Acute, severe infection (e.g., sepsis and opportunistic infections), or active, chronic or persistent infection that might worsen with immunosuppressive treatment (e.g., herpes zoster).
11. Positive serological test for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C serology.
12. Confirmed current active tuberculosis (TB)
13. Central nervous system (CNS) or meningeal involvement, or cord compression by the lymphoma; history of CNS lymphoma
14. History of a severe allergic reaction or anaphylactic reaction to a biological agent or history of hypersensitivity to any component of the trial drug (e.g., hypersensitivity or allergy to murine products).
15. Patients who have significant cardiac disease, including but not limited to history of congestive heart failure (New York Heart Association Class III/IV; see Appendix 7), unstable angina, or uncontrolled cardiac arrhythmia.
16. Uncontrolled or severe hypertension, or cerebrovascular disease.
17. Serious underlying medical conditions that, per the Investigator's discretion, could impair the ability of the patient to participate in the trial
18. Any other co-existing medical or psychological condition(s) that will preclude participation in the study or compromise ability to give informed consent and/or comply with study procedures.
19. Treatment with any investigational medicinal product (IMP) within 4 weeks prior to initiation of 1st infusion of study drug, or treatment with a drug that has not received regulatory approval for any indication within 4 weeks or a minimum of 5 half-lives, whichever is longer, of the 1st infusion of study drug.
20. Receipt of a live/attenuated vaccine within 6 weeks prior to the screening visit.
21. Females who are pregnant, breastfeeding, or planning a pregnancy during the treatment period or within 12 months after the last infusion of study drug.
22. Patients who are investigational site staff members directly involved in the conduct of the trial, and their family members, site staff members otherwise supervised by the investigator, or patients who are Archigen employees directly involved in the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- Research site, Whittier, California, United States
- Research Site, Canberra, Australian Capital Territory, Australia
- Research site, Temuco, Región de la Araucanía, Chile
- Czechia (3):
  - Research site, Hradec Králové
  - Research site, Prague
  - Reasearch site, Prague
- France (2):
  - Research site, Libourne, Gironde
  - Research site, Poitiers, Vienne
- Research site, Hamburg, Germany
- Research site, Budapest, Hungary
- Italy (2):
  - Research site, San Giovanni Rotondo, Foggia
  - Research site, Terni
- Research site, Mexico City, Mexico City, Mexico
- Research site, Pretoria, Gauteng, South Africa
- South Korea (2):
  - Research site, Busan
  - Research site, Seoul
- Spain (3):
  - Research site, L'Hospitalet de Llobregat, Barcelona
  - Research site, Cadiz
  - Research site, Madrid
- Turkey (Türkiye) (4):
  - Research site, Ankara
  - Research site, Istanbul
  - Research site, Mersin
  - Research site, Samsun
- Research site, Norwich, Norfolk, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and one study centres in 29 countries participated in the study. The first participant was enrolled into the study on the 18 January 2017 and the last participant completed week 28 (primary analysis cut-off) on the 17 July 2019.
Pre-assignment Details: A total of 455 participants were consented for the study and 315 participants were randomized in a 1:1 ration to receive SAIT101 (n=157) versus MabThera (n=158).
Groups:
- SAIT101: SAIT101: Dose of 375 mg/m2 body surface area (BSA) intravenous on Weeks 1, 2, 3 and 4,
- MabThera: MabThera: Dose of 375 mg/m2 body surface area (BSA) intravenous on Weeks 1, 2, 3, and 4.
Period: Overall Study
Arm/Group | SAIT101 | MabThera
Started | 157 | 158
Completed Treatment (Received at least one infusion of study drug.) | 156 | 156
Completed (Completed Week 28 (Primary Analysis cut-off)) | 150 | 152
Not Completed | 7 | 6
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Disease Progression | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- SAIT101: SAIT101: Dose of 375 mg/m2 body surface area (BSA) intravenous on Weeks 1, 2, 3, and 4.
- MabThera: MabThera: Dose of 375 mg/m2 body surface area (BSA) intravenous on Weeks 1, 2, 3 and 4.
- Total: Total of all reporting groups
Arm/Group | SAIT101 | MabThera | Total
Number analyzed (Participants) | 157 | 158 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (12.38) | 58.4 (12.78) | 58.1 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 88 | 174
  Male | 71 | 70 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 18
  Not Hispanic or Latino | 136 | 139 | 275
  Unknown or Not Reported | 10 | 12 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 31 | 30 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 115 | 111 | 226
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 8 | 13 | 21
Region of Enrollment [Number; unit: participants]
  Hungary | 4 | 9 | 13
  Czechia | 26 | 24 | 50
  United States | 2 | 3 | 5
  United Kingdom | 3 | 1 | 4
  Spain | 18 | 22 | 40
  South Korea | 10 | 12 | 22
  Turkey | 9 | 9 | 18
  Italy | 13 | 8 | 21
  Mexico | 1 | 1 | 2
  South Africa | 6 | 2 | 8
  Australia | 3 | 5 | 8
  Chile | 2 | 1 | 3
  France | 7 | 8 | 15
  Germany | 5 | 4 | 9
  Ukraine | 5 | 8 | 13
  Thailand | 3 | 1 | 4
  Serbia | 1 | 3 | 4
  Panama | 1 | 0 | 1
  India | 16 | 16 | 32
  Georgia | 2 | 2 | 4
  Guatemala | 2 | 3 | 5
  Belarus | 10 | 5 | 15
  Croatia | 0 | 2 | 2
  Egypt | 7 | 8 | 15
  Philippines | 1 | 1 | 2
Height (cm) [Mean (Standard Deviation); unit: cm] | 165.96 (9.436) | 165.71 (10.650) | 165.84 (10.048)
Weight at baseline (kg) [Mean (Standard Deviation); unit: kg] | 73.80 (15.107) | 73.54 (16.602) | 73.67 (15.850)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.76 (4.857) | 26.66 (4.967) | 26.71 (4.905)
Body Surface Area (m^2) [Mean (Standard Deviation); unit: m^2] | 1.812 (0.2032) | 1.807 (0.2332) | 1.810 (0.2184)
Disease Duration (Years) [Mean (Standard Deviation); unit: years] — Disease duration was derived from initial disease diagnosis date to the date of informed consent. Note that initial disease diagnosis can be confirmed by biopsy after informed consent.
  years | 0.937 (2.1528) | 0.934 (2.5793) | 0.935 (2.3726)
Females of childbearing potential [Count of Participants; unit: Participants] | 24 | 20 | 44
Eastern Co-operative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — The ECOG score is used in the evaluation of cancer patients and can help with prognosis and management of the malignant condition because performance status is highly correlated with survival. A higher ECOG rating score generally equates to a worst outcome. ECOG scores 0 and 1 are defined as:
  ECOG Score 0: Asymptomatic (Fully active, able to carry on all pre-disease activities without restriction);
  ECOG Score 1: Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Participants
    ECOG Score 0 | 132 | 118 | 250
    ECOG Score 1 | 25 | 40 | 65
Antidrug Antibody (ADA) Status at Baseline [Count of Participants; unit: Participants]
  Positive | 3 | 2 | 5
  Negative | 138 | 148 | 286
  Not available | 16 | 8 | 24
Ann Arbor Staging [Count of Participants; unit: Participants] — Ann Arbor staging is the staging system for lymphomas, both in Hodgkin's lymphoma and non-Hodgkin lymphoma.
  Stage I indicates that the cancer is located in a single region.
  Stage II indicates that the cancer is located in two separate regions, an affected lymph node or lymphatic organ and a second affected area.
  Stage III indicates that the cancer has spread to both sides of the diaphragm.
  Stage IV indicates diffuse or disseminated involvement of one or more extralymphatic organs.
  Participants
    Stage I | 1 | 0 | 1
    Stage II | 39 | 37 | 76
    Stage III | 72 | 69 | 141
    Stage IV | 45 | 52 | 97
Type of Ann Arbor Staging [Count of Participants; unit: Participants] — Ann Arbor staging is the staging system for lymphomas, both in Hodgkin's lymphoma (formerly designated Hodgkin's disease) and non-Hodgkin lymphoma (abbreviated NHL). It was initially developed for Hodgkin's, but has some use in NHL. It has roughly the same function as TNM staging in solid tumors
  Ann Arbor Clinical Stage (CS) as obtained by doctor's examination and tests, An Arbor Pathological Stage (PS) as obtained by exploratory laparotomy with splenectomy.
  Participants
    Clinical Stage (CS) | 144 | 140 | 284
    Pathological Stage (PS) | 13 | 18 | 31
Risk Groups According to Follicular Lymphoma International Prognostic Index (FLIP-2) Score [Count of Participants; unit: Participants] — Follicular Lymphoma International Prognostic Index (FLIPI) score of 0 to 1 is considered "low risk" with a 10 year overall survival of 70%. A score of 2 is considered "intermediate risk" with a 10 year overall survival of 50%. Finally, a score of ≥ 3 is considered "high risk" with a 10 year overall survival of 35%.
  Participants
    Low Risk (0 to 1 risk factors) | 102 | 103 | 205
    Intermediate Risk (2 risk factors) | 40 | 41 | 81
    High Risk (Greater than or equal to 3 risk factor | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) at Week 28
Description: Overall Response Rate (ORR) (Complete Response [CR] + Partial Response [PR]) at Week 28, as defined by International Working Group (IWG) criteria 2007. Tumour assessments were assessed by central imaging review per International Working Group (IWG) Criteria 2007. The 95% CI for overall response rate (ORR) was calculated using the Exact method and combined using the Rubin's rule when multiple imputation was applicable.
Time Frame: Baseline (Day 0) to Week 28.
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
percentage of participants | 66.3 [58.64 to 73.87] | 70.6 [63.21 to 77.97]
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Adjusted Difference Rate (%) in Overall Response Rate (ORR) of SAIT101 versus MabThera at Week 28; Test type: Other — The 95%CI (confidence interval) for the difference in the overall response rate (ORR) was calculated using the Newcombe-Wilson method based on CMH (Cochran-Mantel-Haenszel) weight with stratification factor FLIPI-2 (low, intermediate and high risk); Adjusted Difference Rate (%) = -4.2, 95% CI 2-sided [-14.80 to 6.35], Standard Error of Mean 5.40 — Comparison: SAIT101 versus MabThera

2. Secondary Outcome: Overall Response Rate (ORR) at Week 12
Description: Overall Response Rate (ORR) = Complete Response (CR) + Partial Response (PR). Tumour assessments were assessed by central imaging review per the International Working Group (IWG) Criteria 2007. The 95% CI for overall response rate (ORR) was calculated using the Exact method and combined using the Rubin's rule when multiple imputation was applicable.
Time Frame: Baseline (Day 0) to Week 12
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
percentage of participants | 59.6 [51.16 to 67.62] | 70.0 [61.99 to 77.20]
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Adjusted Difference Rate of Overall Response Rate (ORR) of SAIT101 versus MabThera at Week 12; Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted Difference Rate = -10.3, 95% CI 2-sided [-20.92 to 0.61], Standard Error of Mean 5.42 — Comparison: SAIT101 versus MabThera

3. Secondary Outcome: Complete Response (CR) at Weeks 12 and 28
Description: Efficacy Endpoint: Complete Response (CR) at Weeks 12 and 28. Tumour assessments were assessed by central imaging review per International Working Group (IWG) Criteria 2007.
Time Frame: Baseline (Day 0) to Week 12 and Week 28.
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
Participants
  CR at Week 12: number analyzed (Participants) | 145 | 148
  CR at Week 12 | 39 | 37
  CR at Week 28: number analyzed (Participants) | 145 | 144
  CR at Week 28 | 51 | 50

4. Secondary Outcome: Partial Response (PR) at Weeks 12 and 28
Description: Efficacy Endpoint: Partial Response (PR) at Weeks 12 and 28. Tumour assessments were assessed by central imaging review per International Working Group (IWG) Criteria 2007.
Time Frame: Baseline (Day 0) to Week 12 and Week 28.
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
Participants
  PR at Week 12: number analyzed (Participants) | 145 | 148
  PR at Week 12 | 48 | 68
  PR at Week 28: number analyzed (Participants) | 145 | 144
  PR at Week 28 | 47 | 53

5. Secondary Outcome: Stable Disease (SD) at Weeks 12 and 28
Description: Efficacy endpoint: number of participants with Stable Disease (SD) at Weeks 12 and 28. Tumour assessments were assessed by central imaging review per International Working Group (IWG) Criteria 2007.
Time Frame: Baseline (Day 0) to Week 12 and Week 28.
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
Participants
  SD at Week 12: number analyzed (Participants) | 145 | 148
  SD at Week 12 | 50 | 39
  SD at Week 28: number analyzed (Participants) | 145 | 144
  SD at Week 28 | 22 | 27

6. Secondary Outcome: Progressive Disease (PD) at 12 and 28 Weeks
Description: Efficacy endpoint: number of participants with Progressive Disease (PD) at 12 and 28 Weeks. Tumour assessments were assessed by central imaging review per International Working Group (IWG) Criteria 2007.
Time Frame: Baseline (Week 0)to Week 12 and Week 28.
Population: Full Analysis Dataset (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
Participants
  PD at Week 12: number analyzed (Participants) | 145 | 148
  PD at Week 12 | 4 | 1
  PD at Week 28: number analyzed (Participants) | 145 | 144
  PD at Week 28 | 20 | 11

7. Secondary Outcome: Time to Event (TTE)
Description: Time to Event (TTE) is defined as the time of randomisation to the date when an event occurred for a maximum follow-up period of 32 weeks from baseline; an event is disease progression, death due to any cause, or the start of new treatment for follicular lymphoma, whichever comes first.
Time Frame: Baseline (Day 0) to time of event or up to a maximum of 32 weeks, whichever is sooner
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
Weeks | 23.50 (7.500) | 24.08 (6.767)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Time to Event (TTE) Hazard Ratio (HR) of SAIT101:MabThera. The TTE is defined as the time from the date of randomization to the date when an event occurs; an event is disease progression as assessed by Investigator, death due to any cause, or the start of new treatment, whichever comes first; Test type: Other — The estimated Hazard Ratio with 95% CI was obtained from Cox regression model; however, stratification factors, ie, FLIPI-2 (low, intermediate and high risk), were only taken into account if FLIPI-2 score=all; Hazard Ratio (HR) = 1.724, 95% CI 2-sided [0.853 to 3.482] — Hazard Ration of TTE SAIT101:MabThera

8. Other Pre Specified Outcome: Truncated Area Under the Concentration-time Curve (AUC) Over the First and Fourth Dosing Intervals (AUC0 168,w1, AUC0-168,w4).
Description: Pharmacokinetic endpoint: truncated area under the concentration-time curve (AUC) over the first (Day 1) and fourth (Day 22) dosing intervals (AUC0 168,w1, AUC0-168,w4).
Time Frame: Baseline (Day 0) to dosing on Week 1 and Week 4
Population: Pharmacokinetic Analysis Set (PAS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: H*µg/ml
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 76 | 72
H*µg/ml
  AUC0-168, week 1: number analyzed (Participants) | 60 | 58
  AUC0-168, week 1 | 20140 (18.7) | 19860 (18.3)
  AUC0-168, week 4: number analyzed (Participants) | 53 | 43
  AUC0-168, week 4 | 41290 (19.0) | 42600 (19.4)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Statistical Comparison: geometric least square (GLS) Mean Ratio (90% Confidence Interval (CI)) (%) of SAIT101 versus MabThera Area Under the Concentration time Curve Day 0 to Week 1 (AUC0-168,w1) (h×µg/mL). The statistical comparison of the loge-transformed primary parameters between treatments is based on an analysis of variance model with fixed effect for treatment; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%); GLS Mean Difference (%) = 101.39, 90% CI 2-sided [95.86 to 107.24] — Comparison: SAIT101 versus MabThera. Equivalence was demonstrated for SAIT101 and MabThera with exposure pharmacokinetic parameter AUC0-168,w1 within the standard acceptance limits for bioequivalence (80.00% to 125.00%)
Statistical Analysis 2: Comparison: SAIT101 vs MabThera; Statistical Comparison: geometric least square (GLS) Mean Ratio (90% Confidence Interval (CI)) %) of SAIT101 versus MabThera Area Under the Concentration time Cure Day 0 to Week 4 (AUC0-168,w4) (h×µg/mL). The statistical comparison of the loge-transformed primary parameters between treatments is based on an analysis of variance model with fixed effect for treatment; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%); GLS Mean Difference (%) = 96.92, 90% CI 2-sided [90.85 to 103.40] — Comparison: SAIT101 versus MabThera. Pharmacokinetic equivalence was demonstrated for SAIT101 and MabThera with exposure PK parameter AUC0-168,w4 within the standard acceptance limits for bioequivalence (80.00% to 125.00%)

9. Other Pre Specified Outcome: Maximum Concentration (Cmax) After the First Dose and the Fourth Dose (Cmax,w1, Cmax,w4).
Description: Pharmacokinetic endpoint: maximum plasma concentration (Cmax, µg/ml ) after the first dose (Week 1) and the fourth dose (week 4) (Cmax,w1, Cmax,w4).
Time Frame: Baseline (Day 0) to dosing on Week 1 and Week 4
Population: Pharmacokinetic Analysis Set (PAS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/ml
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 76 | 72
µg/ml
  Cmax, week 1: number analyzed (Participants) | 62 | 62
  Cmax, week 1 | 199.3 (22.1) | 200.6 (27.5)
  Cmax, week 4: number analyzed (Participants) | 62 | 56
  Cmax, week 4 | 333.6 (22.8) | 336.2 (20.2)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Statistical Comparison: geometric least square (GLS) Mean Ratio (90% CI) (%) of SAIT101 versus MabThera maximum plasma concentration at Week 1 (Cmax,w1) (h×µg/mL). The statistical comparison of the loge-transformed primary parameters between treatments is based on an analysis of variance model with fixed effect for treatment; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00; GLS Mean Ratio (%) = 99.35, 90% CI 2-sided [90.85 to 103.40] — Comparison: SAIT101 versus MabThera. Pharmacokinetic equivalence was demonstrated for SAIT101 and MabThera with Cmax,w1 exposure within the standard acceptance limits for bioequivalence (80.00% to 125.00%)
Statistical Analysis 2: Comparison: SAIT101 vs MabThera; Statistical Comparison: geometric least square (GLS) Mean Ratio (90% CI) (%) of SAIT101 versus MabThera maximum plasma concentration at Week 4 (Cmax,w1) (h×µg/mL). The statistical comparison of the loge-transformed primary parameters between treatments is based on an analysis of variance model with fixed effect for treatment; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%); GLS Mean Ration (%) = 99.23, 90% CI 2-sided [92.96 to 105.92] — Comparison: SAIT101 versus MabThera. Pharmacokinetic equivalence was demonstrated for SAIT101 and MabThera with exposure PK parameter Cmax,w4 within the standard acceptance limits for bioequivalence (80.00% to 125.00%)

10. Other Pre Specified Outcome: Accumulation Ratio for AUC0-168 Obtained From the Fourth Dose Versus the First Dose (RAUC).
Description: Pharmacokinetic endpoint: accumulation ratio for the Area Under the Concentration Time Cure 0 to 168 hours (AUC0-168) obtained from the fourth dose (Week 4) versus the first dose (Week 1) (RAUC). Accumulation ratio, calculated for AUC0-168 as (AUC0 168,w4/AUC0 168,w1).
Time Frame: Baseline (Day 0) to dosing on Week 1 and Week 4
Population: Pharmacokinetic Analysis Set (PAS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 76 | 72
Ratio | 2.075 (17.2) | 2.137 (21.0)

11. Other Pre Specified Outcome: Accumulation Ratio for the Maximum Plasma Concentration (Cmax) From the Fourth Dose Versus the First Dose (RCmax).
Description: Pharmacokinetic endpoint: accumulation ratio for maximum plasma (Cmax) ratio from the fourth dose on Week 4 versus the first dose of treatment on Week 1 (RCmax). Accumulation ratio, calculated for Cmax as (Cmax,w4/Cmax,w1).
Time Frame: Baseline (Day 0) to dosing on Week 1 and Week 4
Population: Pharmacokinetic Analysis set (PAS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 76 | 72
Ratio | 1.706 (23.2) | 1.671 (21.0)

12. Other Pre Specified Outcome: Trough Concentrations on Days 1, 8, 15, 22, and 29 (Ctrough).
Description: Pharmacokinetic endpoint: trough plasma concentration (Ctrough) during the dosing phase on Days 1, 8, 15, 22, and 29. Concentrations at predose on Days 8, 15, and 22 (µg/mL) and the time equivalent to the predose on Day 29, obtained directly from the observed concentration versus time data.
Time Frame: Baseline (Day 0) to Days 1, 8, 15, 22 and 29
Population: Pharmacokinetic Analysis Set (PAS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/ml
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 76 | 72
µg/ml
  Ctrough Day 8: number analyzed (Participants) | 74 | 67
  Ctrough Day 8 | 60.60 (45.5) | 61.00 (43.4)
  Ctrough Day 15: number analyzed (Participants) | 67 | 63
  Ctrough Day 15 | 108.1 (26.0) | 107.3 (32.0)
  Ctrough Day 22: number analyzed (Participants) | 71 | 64
  Ctrough Day 22 | 143 (23.8) | 143.3 (30.0)
  Ctrough Day 29: number analyzed (Participants) | 65 | 56
  Ctrough Day 29 | 181.7 (22.1) | 190.4 (26.1)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Statistical Comparison: geometric least square (GLS) Mean Ratio (90% CI) (%) of SAIT101 versus MabThera trough plasma concentration at the end of the dosing period (Day 29) (Ctrough,d29) (µg/mL) . The statistical comparison of the log-transformed primary parameters between treatments is based on an analysis of variance model with fixed effect for treatment; Test type: Equivalence — Standard acceptance limits for bioequivalence (80.00% to 125.00%); GLS Mean Ratio (%) = 95.45, 90% CI 2-sided [88.85 to 102.55] — Comparison: SAIT101 versus MabThera. Pharmacokinetic equivalence was demonstrated for SAIT101 and MabThera with exposure PK parameter Ctrough,d29 within the standard acceptance limits for bioequivalence (80.00% to 125.00%)

13. Other Pre Specified Outcome: Observed Change From Baseline CD19+ B-Lymphocyte Cluster of Differentiation 19 (CD-19+ B-Cell) Counts up to Week 28
Description: Pharmacodynamic Endpoint: Arithmetic mean observed change from baseline of B-lymphocyte antigen cluster of differentiation 19 (CD-19+ B-cell) counts (cells/μL) up to Week 28 by treatment.
Time Frame: Baseline (Day 1) to Weeks 1, 2, 3, 4, 5, 12, 20 and 28.
Population: Pharmacodynamic Analysis Set (PDS)
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 76 | 72
cells/μL
  Week 1 Mean Change from Baseline: number analyzed (Participants) | 58 | 61
  Week 1 Mean Change from Baseline | -128.0 (115.71) | -141.6 (120.90)
  Week 2 Mean Change from Baseline: number analyzed (Participants) | 60 | 58
  Week 2 Mean Change from Baseline | -144.1 (123.34) | -146.8 (138.76)
  Week 3 Mean Change from Baseline: number analyzed (Participants) | 59 | 54
  Week 3 Mean Change from Baseline | -142.8 (122.63) | -157.4 (102.03)
  Week 4 Mean Change from Baseline: number analyzed (Participants) | 57 | 54
  Week 4 Mean Change from Baseline | -141.5 (122.92) | -141.2 (102.03)
  Week 5 Mean Change from Baseline: number analyzed (Participants) | 63 | 58
  Week 5 Mean Change from Baseline | -140.0 (120.74) | -158.5 (134.27)
  Week 12 Mean Change from Baseline: number analyzed (Participants) | 62 | 56
  Week 12 Mean Change from Baseline | -144.2 (122.09) | -160.1 (134.09)
  Week 20 Mean Change from Baseline: number analyzed (Participants) | 61 | 58
  Week 20 Mean Change from Baseline | -140.8 (117.98) | -159.5 (135.63)
  Week 28 Mean Change from Baseline: number analyzed (Participants) | 60 | 58
  Week 28 Mean Change from Baseline | -136.6 (122.80) | -148.2 (134.79)

14. Other Pre Specified Outcome: Percent Change From Baseline CD19+ B-Lymphocyte Cluster of Differentiation 19 (CD-19+ B-Cell) Counts up to Week 28
Description: Pharmacodynamic Endpoint: percent change from baseline of B-lymphocyte antigen cluster of differentiation 19 (CD-19+ B-cell) counts (cells/μL) up to Week 28 by treatment.
Time Frame: Baseline (Day 1) to Weeks 1, 2, 3, 4, 5, 12, 20 and 28.
Population: Pharmacodynamic Analysis Set (PDS)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 76 | 72
Percent change
  Week 1 % Change from Baseline: number analyzed (Participants) | 58 | 60
  Week 1 % Change from Baseline | -89.02 (26.324) | -95.58 (8.294)
  Week 2 % Change from Baseline: number analyzed (Participants) | 66 | 59
  Week 2 % Change from Baseline | -100.00 (0.000) | -94.62 (1.230)
  Week 3 % Change from Baseline: number analyzed (Participants) | 59 | 57
  Week 3 % Change from Baseline | -100.00 (0.000) | -100.00 (0.000)
  Week 4 % Change from Baseline: number analyzed (Participants) | 57 | 53
  Week 4 % Change from Baseline | -100.00 (0.000) | -100.00 (0.000)
  Week 5 % Change from Baseline: number analyzed (Participants) | 63 | 57
  Week 5 % Change from Baseline | -100.00 (0.000) | -100.00 (0.000)
  Week 12 % Change from Baseline: number analyzed (Participants) | 62 | 55
  Week 12 % Change from Baseline | -100.00 (0.000) | -100.00 (0.000)
  Week 20 % Change from Baseline: number analyzed (Participants) | 61 | 57
  Week 20 % Change from Baseline | -100.00 (0.000) | -100.00 (0.000)
  Week 28 % Change from Baseline: number analyzed (Participants) | 60 | 72
  Week 28 % Change from Baseline | -97.42 (12.749) | -100.00 (0.000)

15. Other Pre Specified Outcome: Area Under the Curve Change From Baseline B-lymphocyte Cluster of Differentiation 19 (CD19+ B-cell) Count Time Curve (AUEC) Over the Dosing Interval
Description: Pharmacodynamic Endpoint: Area under the change from baseline CD19+ B-cell count time curve (AUEC) over the first dosing interval on week 1 from time 0 to the time prior to the second dose (AUEC0 168,w1), AUEC over the second dosing interval on week 2 from time 0 to the time prior to the third dose (AUEC0-168,w2), AUEC over the third dosing interval on week 3 from time 0 to the time prior to the fourth dose (AUEC0-168,w3), AUEC over the fourth dosing interval on week 4 from time 0 to 168 hours post dose (AUEC0-168,w4), AUEC from time 0 on week 1 to the time point on week 12 (AUEC0-w12), AUEC from time 0 on week 1 to the time point on week 28 (AUEC0 w28) for the change from baseline CD19+ B-cell count data.
Time Frame: Baseline (Day 0) to Week 1, 2, 3, 4 12 and 28.
Population: Pharmacodynamic Analysis Set
Measure: Mean (Standard Deviation); unit: cells*day/µL)
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 76 | 72
cells*day/µL)
  AUEC0-168,w1 (cells*day/µL): number analyzed (Participants) | 54 | 59
  AUEC0-168,w1 (cells*day/µL) | -946.0 (830.29) | -1000 (891.82)
  AUEC0-168,w2 (cells*day/µL): number analyzed (Participants) | 58 | 58
  AUEC0-168,w2 (cells*day/µL) | -987.2 (997.57) | -1104 (947.68)
  AUEC0-168,w3 (cells*day/µL): number analyzed (Participants) | 58 | 58
  AUEC0-168,w3 (cells*day/µL) | -944.8 (910.79) | -1073 (930.95)
  AUEC0-168,w4 (cells*day/µL): number analyzed (Participants) | 60 | 56
  AUEC0-168,w4 (cells*day/µL) | -956.3 (728.52) | -1196 (1153.7)
  AUEC0-w12 (cells*day/µL): number analyzed (Participants) | 62 | 60
  AUEC0-w12 (cells*day/µL) | 11330 (9854.1) | -12280 (10185)
  AUEC0-w28 (cells*day/µL): number analyzed (Participants) | 60 | 58
  AUEC0-w28 (cells*day/µL) | -26370 (22794) | -28860 (25439)

16. Other Pre Specified Outcome: Normalized Area Under the Curve Change From Baseline B-lymphocyte Cluster of Differentiation 19 (CD19+ B-cell) Count Time Curve (AUEC) Over the Dosing Interval
Description: Pharmacodynamic Endpoint: Area under the change from baseline CD19+ B-cell count time curve (AUEC) over the first dosing interval on week 1 from time 0 to the time prior to the second dose (AUEC0 168,w1), AUEC over the second dosing interval on week 2 from time 0 to the time prior to the third dose (AUEC0-168,w2), AUEC over the third dosing interval on week 3 from time 0 to the time prior to the fourth dose (AUEC0-168,w3), AUEC over the fourth dosing interval on week 4 from time 0 to 168 hours post dose (AUEC0-168,w4), AUEC from time 0 on week 1 to the time point on week 12 (AUEC0-w12), AUEC from time 0 on week 1 to the time point on week 28 (AUEC0 w28) for the change from baseline CD19+ B-cell count data. The time-normalized AUEC parameters presented were calculated by dividing the respective AUEC by the time interval used to calculate the AUEC.
Time Frame: Baseline (Day 0) to Week 1, 2, 3, 4 12 and 28.
Population: Pharmacodynamic Analysis Set
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 76 | 72
cells/µL
  AUEC0-168,w1, normalized (cells/µL) | -135.0 (118.88) | -142.1 (125.23)
  AUEC0-168,w2, normalized (cells/µL): number analyzed (Participants) | 58 | 58
  AUEC0-168,w2, normalized (cells/µL) | -137.1 (123.43) | -155.1 (133.38)
  AUEC0-168,w3, normalized (cells/µL): number analyzed (Participants) | 58 | 58
  AUEC0-168,w3, normalized (cells/µL) | -134.3 (121.75) | -155.7 (135.47)
  AUEC0-168,w4, normalized (cells/µL): number analyzed (Participants) | 60 | 56
  AUEC0-168,w4, normalized (cells/µL) | -138.7 (121.62) | -159.2 (136.55)
  AUEC0-w12, normalized (cells/µL): number analyzed (Participants) | 62 | 56
  AUEC0-w12, normalized (cells/µL) | -143.0 (121.38) | -158.7 (133.02)
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Statistical Comparison of CD19+ B-cell Pharmacodynamic Parameters (Pharmacodynamic Analysis Set). Area under the pharmacodynamic time effect curve from baseline (Time 0) to Week 1 (AUEC0-168,w1), normalized (cells/µL). The statistical comparison of the between treatments is based on an analysis of covariance (ANOVA) model with fixed effect for treatment and a covariate for baseline value; Test type: Other; Mean Difference (Final Values) = 7.2, 90% CI 2-sided [-31.0 to 45.4] — Comparison: SAIT101 versus MabThera
Statistical Analysis 2: Comparison: SAIT101 vs MabThera; Statistical Comparison of CD19+ B-cell Pharmacodynamic Parameters (Pharmacodynamic Analysis Set). Area under the pharmacodynamic time effect curve from baseline (Time 0) to Week 2 (AUEC0-168,w2), normalized (cells/µL). The statistical comparison of the between treatments is based on an analysis of covariance (ANOVA) model with fixed effect for treatment and a covariate for baseline value; Test type: Other; Mean Difference (Final Values) = 18.0, 90% CI 2-sided [-21.6 to 57.6] — Comparison: SAIT101 versus MabThera
Statistical Analysis 3: Comparison: SAIT101 vs MabThera; Statistical Comparison of CD19+ B-cell Pharmacodynamic Parameters (Pharmacodynamic Analysis Set). Area under the pharmacodynamic time effect curve from baseline (Time 0) to Week 3 (AUEC0-168,w3), normalized (cells/µL). The statistical comparison of the between treatments is based on an analysis of covariance (ANOVA) model with fixed effect for treatment and a covariate for baseline value; Test type: Other; Mean Difference (Final Values) = 21.4, 90% CI 2-sided [-18.3 to 61.0] — Comparison: SAIT101 versus MabThera
Statistical Analysis 4: Comparison: SAIT101 vs MabThera; Statistical Comparison of CD19+ B-cell Pharmacodynamic Parameters (Pharmacodynamic Analysis Set). Area under the pharmacodynamic time effect curve from baseline (Time 0) to Week 4 (AUEC0-168,w4), normalized (cells/µL). The statistical comparison of the between treatments is based on an analysis of covariance (ANOVA) model with fixed effect for treatment and a covariate for baseline value; Test type: Other; Mean Difference (Final Values) = 20.4, 90% CI 2-sided [-19.3 to 60.2] — comparison: SAIT101 versus MabThera
Statistical Analysis 5: Comparison: SAIT101 vs MabThera; Statistical Comparison of CD19+ B-cell Pharmacodynamic Parameters (Pharmacodynamic Analysis Set). Area under the pharmacodynamic time effect curve from baseline (Time 0) to Week 12 (AUEC0-168,w12), normalized (cells/µL). The statistical comparison of the between treatments is based on an analysis of covariance (ANOVA) model with fixed effect for treatment and a covariate for baseline value; Test type: Other; Mean Difference (Final Values) = 15.7, 90% CI 2-sided [-23.1 to 54.6] — Comparison: SAIT101 versus MabThera
Statistical Analysis 6: Comparison: SAIT101 vs MabThera; Statistical Comparison of CD19+ B-cell Pharmacodynamic Parameters (Pharmacodynamic Analysis Set). Area under the pharmacodynamic time effect curve from baseline (Time 0) to Week 28 (AUEC0-168,w28), normalized (cells/µL). The statistical comparison of the between treatments is based on an analysis of covariance (ANOVA) model with fixed effect for treatment and a covariate for baseline value; Test type: Other; Mean Difference (Final Values) = 12.8, 90% CI 2-sided [-26.0 to 51.8] — Comparison: SAIT101 versus MabThera

17. Other Pre Specified Outcome: Incidence of Antidrug Antibodies (ADA) and Neutralising Antibody (NAb) by Visit
Description: Immunogenicity endpoint: incidence of antidrug antibodies (ADA) and Neutralising Antibody (NAb). Immunogenicity sampling was performed pre-dose at Day 1, weeks 2, 3 and 4 and at any time during the visits at weeks 5, 12, 20 and 28.
Time Frame: Pre-dose on Day 1 to Weeks 5, 12, 20 and 28.
Population: Safety Analysis Set (SAS
Measure: Count of Participants; unit: Participants
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 152 | 156
Participants
  Week 1 (Baseline) ADA: number analyzed (Participants) | 141 | 150
  Week 1 (Baseline) ADA: Negative | 138 | 148
  Week 1 (Baseline) ADA: Positive | 3 | 2
  Week 1 (Baseline) NAb: number analyzed (Participants) | 3 | 2
  Week 1 (Baseline) NAb: Negative | 3 | 2
  Week 1 (Baseline) NAb: Positive | 0 | 0
  Week 2 ADA: number analyzed (Participants) | 144 | 152
  Week 2 ADA: Negative | 143 | 152
  Week 2 ADA: Positive | 1 | 0
  Week 2 NAb: number analyzed (Participants) | 1 | 0
  Week 2 NAb: Negative | 1 | 0
  Week 2 NAb: Positive | 0 | 0
  Week 3 ADA: number analyzed (Participants) | 143 | 150
  Week 3 ADA: Negative | 138 | 148
  Week 3 ADA: Positive | 5 | 2
  Week 3 NAb: number analyzed (Participants) | 5 | 2
  Week 3 NAb: Negative | 5 | 2
  Week 3 NAb: Positive | 0 | 0
  Week 4 ADA: number analyzed (Participants) | 147 | 149
  Week 4 ADA: Negative | 145 | 149
  Week 4 ADA: Positive | 2 | 0
  Week 4 NAb: number analyzed (Participants) | 2 | 0
  Week 4 NAb: Negative | 2 | 0
  Week 4 NAb: Positive | 0 | 0
  Week 5 ADA: number analyzed (Participants) | 141 | 145
  Week 5 ADA: Negative | 139 | 145
  Week 5 ADA: Positive | 2 | 0
  Week 5 NAb: number analyzed (Participants) | 2 | 0
  Week 5 NAb: Negative | 2 | 0
  Week 5 NAb: Positive | 0 | 0
  Week 12 ADA: number analyzed (Participants) | 140 | 144
  Week 12 ADA: Negative | 137 | 144
  Week 12 ADA: Positive | 3 | 0
  Week 12 NAb: number analyzed (Participants) | 3 | 0
  Week 12 NAb: Negative | 3 | 0
  Week 12 NAb: Positive | 0 | 0
  Week 20 ADA: number analyzed (Participants) | 138 | 148
  Week 20 ADA: Negative | 131 | 144
  Week 20 ADA: Positive | 7 | 4
  Week 20 NAb: number analyzed (Participants) | 7 | 4
  Week 20 NAb: Negative | 7 | 4
  Week 20 NAb: Positive | 0 | 0
  Week 28 ADA: number analyzed (Participants) | 136 | 145
  Week 28 ADA: Negative | 126 | 129
  Week 28 ADA: Positive | 10 | 16
  Week 29 NAb: number analyzed (Participants) | 10 | 16
  Week 29 NAb: Negative | 9 | 16
  Week 29 NAb: Positive | 1 | 0

18. Other Pre Specified Outcome: Observed Change From Baseline for Immunoglobulins G and M by Scheduled Time
Description: Exploratory pharmacodynamic endpoint: Mean (SD) Change from Baseline of Immunoglobulin (IgG) and immunoglobulin M (IgM) (mg/dL) by Scheduled Time for Each Treatment (Safety Analysis Set). Samples for IgG and IgM assessment were collected at Baseline and Weeks 1, 2, 3, 4, 5, 12, 20 and 28.
Time Frame: Baseline to Weeks 1, 2, 3, 4, 5, 12, 20 and 28.
Population: Safety Analysis Set (SAS)
Measure: Mean (Standard Deviation); unit: Mg/dL
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
Mg/dL
  IgG Week 2 | -0.21 (132.687) | -14.79 (132.64)
  IgG Week 3 | -17.08 (157.848) | -30.04 (124.814)
  IgG Week 4 | -36.31 (132.326) | -34.64 (156.790)
  IgG Week 5 | -34.62 (162.748) | -38.21 (170.758)
  IgG Week 12 | -28.15 (159.898) | -2.30 (202.017)
  IgG Week 20 | -26.86 (189.937) | -22.40 (173.420)
  IgG Week 28 | -19.33 (200.69) | 8.70 (238.309)
  IgM Week 2 | 0.34 (18.018) | 4.60 (28.273)
  IgM Week 3 | 0.87 (25.092) | 2.12 (32.569)
  IgM Week 4 | 0.64 (31.836) | 0.03 (30.009)
  IgM Week 5 | -1.91 (29.521) | -2.02 (21.651)
  IgM Week 12 | 8.02 (37.876) | 9.12 (21.671)
  IgM Week 20 | -12.94 (46.966) | -14.35 (26.012)
  IgM Week 28 | -22.08 (29.200) | -20.85 (37.475)

19. Other Pre Specified Outcome: Exploratory Analyses of Tumor Response and Time to Event
Description: Exploratory Efficacy Endpoint: Analyses of Tumor Response and Time to Event, as Determined by the Combined International Working Group (IWG) Criteria 2014, Lugano Classification and IWG Criteria 2007 (Central Assessment) (Full Analysis Set)
Time Frame: Baseline (Day 0) to Week 28
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
Participants
  Complete Response (CR): number analyzed (Participants) | 145 | 144
  Complete Response (CR) | 53 | 50
  Partial Response (PR): number analyzed (Participants) | 145 | 144
  Partial Response (PR) | 47 | 55
  Stable Disease (SD): number analyzed (Participants) | 145 | 144
  Stable Disease (SD) | 21 | 25
  Progressive Disease (PD): number analyzed (Participants) | 145 | 144
  Progressive Disease (PD) | 19 | 11
  Unknown (UKN): number analyzed (Participants) | 145 | 144
  Unknown (UKN) | 1 | 2
  No Evidence of Disease (NED): number analyzed (Participants) | 145 | 144
  No Evidence of Disease (NED) | 4 | 1

20. Other Pre Specified Outcome: Subgroups and Treatment Interactions of Overall Response Rate (ORR) by Region, Age, Gender and Anti-Drug Antibody (ADA) Status at Week 28.
Description: Exploratory Efficacy Endpoint: Overall Response Rate (ORR) at Week 28 by Region, Age, Gender and Anti-Drug antibody (ADA) status. ADA status through Week 28 is 'Positive' if 'Positive' at any time point, and 'Negative' if 'Negative' at all time points. The 95% CI (confidence interval) for overall response rate (ORR) was calculated using the Exact method. The results presented in this table are based on the non-responder imputed data.
Time Frame: Baseline (Day 0) to Week 28
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SAIT101 | MabThera
Number analyzed (Participants) | 157 | 158
percentage of participants
  ORR European Union (%) | 68.5 [57.96 to 77.77] | 70.2 [59.90 to 79.21]
  ORR Other Region (%) | 54.8 [41.03 to 66.30] | 57.8 [44.82 to 70.06]
  ORR Age 10-60 years (%) | 58.6 [47.55 to 69.08] | 70.6 [59.71 to 99.98]
  ORR Age >60 years (%) | 67.1 [54.88 to 77.91] | 58.9 [46.77 to 70.29]
  ORR Gender Female (%) | 72.1 [61.38 to 81.23] | 67.0 [56.21 to 76.70]
  ORR Gender Male (%) | 50.7 [38.56 to 62.78] | 62.9 [50.48 to 74.11]
  ORR ADA Positive (%) | 42.1 [20.25 to 66.50] | 57.1 [34.02 to 78.18]
  ORR ADA Negative (%) | 65.4 [56.68 to 73.44] | 66.7 [58.04 to 74.54]
Statistical Analysis 1: Comparison: SAIT101 vs MabThera; Exploratory statistical analysis: Comparison of Overall Response Rate (ORR) by Region (European Union / Other). The interaction p-value for the Region subgroup was calculated based upon the full set of data, and based on a Cochran Mantel Haenszel (CMH) model including treatment, and applicable stratification covariate; Test type: Other; p = 0.587, Gail-Simon — The p-value was calculated using Gail-Simon Test for Qualitative Interactions
Statistical Analysis 2: Comparison: SAIT101 vs MabThera; Exploratory statistical analysis. Overall Response Rate by Age Group (18-60 years and >60 years). The interaction p-value for the Age subgroup was calculated based upon the full set of data, and based on a Cochran Mantel Haenszel (CMH) model including treatment, and applicable stratification covariate; Test type: Other; p = 0.421, Gail-Simon — The p-value was calculated using Gail-Simon Test for Qualitative Interactions
Statistical Analysis 3: Comparison: SAIT101 vs MabThera; Exploratory statistical analysis. Comparison of Overall Response Rate (ORR) by Gender (Male / Female). The interaction p-value for the Gender subgroup was calculated based upon the full set of data, and based on a Cochran Mantel Haenszel (CMH) model including treatment, and applicable stratification covariate. The p-value was calculated using Gail-Simon Test for Qualitative Interactions; Test type: Other; p = 0.288, Gail-Simon — The p-value was calculated using Gail-Simon Test for Qualitative Interactions
Statistical Analysis 4: Comparison: SAIT101 vs MabThera; Exploratory statistical analysis. Comparison of Overall Response Rate (ORR) by Anti-drug Antibody (ADA) status (Positive / Negative). The interaction p-value for the ADA subgroup was calculated based upon the full set of data, and based on a Cochran Mantel Haenszel (CMH) model including treatment, and applicable stratification covariate; Test type: Other; p = 0.588, Gail-Wilson — The p-value was calculated using Gail-Simon Test for Qualitative Interactions

ADVERSE EVENTS:
Time Frame: After the participant signed the Informed Consent Form (ICF), but prior to the initiation of study drug, only Serious Adverse Events (SAEs) caused by a protocol mandated procedure should be reported (e.g. SAEs related to invasive procedures such as biopsies). All adverse events were collected for each patient from the start of the first infusion of study drug on Day 1 until the Week 28 Data-cut off.
Description: All AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) v22.1. If an AE changed from non-SAE to be an SAE, it was treated as a new event and was counted as 2 events in the AE summary. A treatment-emergent AE (TEAE) was defined as any AE with an onset date on or after the date of the first dose of study treatment until Week 28, or the End of Study (EOS) visit, if earlier.
Arm/Group | SAIT101 | MabThera
All-Cause Mortality (participants affected / at risk) | 0/157 | 1/158
Serious Adverse Events (participants affected / at risk) | 3/157 | 4/158
Other Adverse Events (participants affected / at risk) | 85/157 | 70/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAIT101 (N=157) | MabThera (N=158)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Cystitis klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAIT101 (N=157) | MabThera (N=158)
Neutrpopenia (Blood and lymphatic system disorders) | 7 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5)
Fatigue (General disorders) | 6 (7) | 7 (11)
Asthenia (General disorders) | 4 (4) | 4 (4)
Pyrexia (General disorders) | 4 (4) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 18 (27) | 26 (30)
Alanine aminotransferase increased (Investigations) | 3 (4) | 4 (4)
Headache (Nervous system disorders) | 9 (10) | 2 (5)
Paraesthesia (Nervous system disorders) | 4 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 8 (8)
Hypertension (Vascular disorders) | 4 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT02809053/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT02809053/SAP_001.pdf